CLINICAL TRIAL: NCT04420013
Title: Colorectal Cancer Immunomodulation Combined to Radiofrequency ablatIon
Brief Title: Colorectal Cancer Immunomonitoring Combined With Radiofrequency ablatIon
Acronym: ColIBRI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 19RME-ColIBRI
Record Dates: First submitted 2020-05-28; First posted 2020-06-09 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-07

CONDITIONS: Colorectal Cancer; Radiofrequency ablatIon
Keywords: colorectal cancer; immunomonitoring; radiofrequency ablatIon
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Standard plasma sampling (15 ml) as usual care, with the following timeframe:
  * preoperative (baseline);
  * at 24 hours post-operative;
  * at 2 months post-operative.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- exposed group: for CRC patients with non-resectable hepatic metastases: surgery for CRC combined with RFA.
- no-exposed group: for CRC patients with resectable metastases: surgery only without RFA.

SUMMARY:
The primary objective of the study aims to compare soluble CD154 (CD40L) levels before and after radiofrequency ablation (RFA) in patients with colorectal cancer (CRC) liver metastases.

The secondary objectives aims:

* to compare soluble CD154 (sCD40-L) levels before and after treatment by RFA or surgery alone in patients with CRC liver metastases;
* to study the feasibility and reliability of soluble CD154 (sCD40-L) levels to detect and quantify the induction of immun response in CRC liver metastases patients after RFA;
* to study the impact of surgery on plasma soluble CD154 levels;
* to study association between CD154 expression level before and after RFA in CRC liver metastases patients and relapses rate at 1 year.

DETAILED DESCRIPTION:
Radiofrequency ablation (RFA) of colorectal liver metastases activates a specific T-cell response that is ineffective in avoiding recurrence. Local immunomodulation garnered interests as a way to improve the immune response. It was interesting in improving the RFA immune response priming to propose a curative treatment of colorectal cancer (CRC) based on antitumor immunity. Early study of the investigators demonstrated that the RFA did not increase the tumor infiltrating lymphocytes in secondary distant tumors of patients and in mice model and could not avoid relapse. The lack of an effective distant immune response in patients treated with RFA confirmed the relevance of the combination strategy.

Another study on the predictive value of cytokines/chemokines in rectal cancer (RC) patients receiving chemoradiation therapy (CRT) demonstrate that, the pre-CRT levels of soluble CD40-ligand (sCD40L) and the post-CRT levels of chemokine ligand-5 (CCL-5) were significantly associated with the depth of tumor invasion and with venous invasion. A significant correlation between pre-CRT platelet counts and sCD40L was observed in patients with a favorable response.

Today there is no validated biomarker for the indication of immunotherapy after local treatment on metastases of colorectal cancer.

This is a prospective, monocentric study which will be realized with the routine care and usual management. There will be any added intervention for enrolled patients during the study. All eligible patients will be enrolled and followed in the Department of digestive surgery of Ambroise Paré Hospital - APHP.

The duration of enrollment will last 6 months. The duration of follow-up for each patient will be up to 12 month.

Data collection: the medical data will be collected and recorded by Doctor Malafosse in a Excel file.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven CRC;
2. Age ≥ 18 years;
3. For group of ablation by radiofrequency: non-resectable liver metastases from CRC without detectable extra-hepatic disease, on abdomino-pelvic computed tomography (CT) or magnetic resonance imaging (MRI) and chest CT by the consulting hepatobiliary surgeon and radiologist.
4. For surgery group: only histologically proven CRC or treatable resectable liver metastases by only surgery without radiofrequency;
5. Metastatic involvement of the liver ≤50%;
6. Complete treatment of all liver lesions judged possible, either by RFA alone or by combination with resection of resectable lesions and RFA of the remaining non-resectable liver deposits;
7. Serum albumin ≥ 30 g / L ;
8. White blood cell count (WBC) ≥ 3 000 / ml;
9. Absolute lymphocytes count ≥ 1000 / ml;
10. Registration in a national health care system included CMU;
11. Any other prior therapy directed at the malignant tumor, including chemotherapy; chemoembolization therapy, molecular targeted therapy (including antiangiogenics), and radiotherapy, must be discontinued at least 3 weeks before day 1 on trial.

Exclusion Criteria:

1. Major surgical procedures within 28 days before RFA;
2. Receipt of the last dose of anticancer therapy (investigational product, chemotherapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies) ≤ 21 days prior to the RFA;
3. Histology other than adenocarcinoma;
4. Hilar lymph node or pedicular metastases;
5. Obstructive jaundice (bilirubin > 1.5 ULN) without adequate biliary drainage;
6. Any unresolved toxicity NCI CTCAE Grade ≥ 2 from previous anticancer therapy with the exception of alopecia, neuropathy, and the laboratory values defined in the inclusion criteria;
7. History of allogenic organ transplantation;
8. Any systemic steroid therapy whatever the duration of this corticotherapy;

   Note: The following are exceptions to this criterion:
   * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
   * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication);
9. Active infection including tuberculosis, hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies); Note: Patients with past HBV infection or resolved HBV infection (defined as having a negative HBsAg test and a positive hepatitis B core antigen [HBc] antibody test) are eligible.

   Note: Patients positive for HCV antibody are eligible only if polymerase chain reaction testing is negative for HCV ribonucleic acid (RNA).
10. Diagnosis of any second malignancy within the last 5 years, except for adequately treated basal cell or squamous cell skin cancer, or in situ carcinoma of the cervix uteri;
11. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]), that has required systemic treatment (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); Note: Patients with vitiligo, alopecia, or any chronic skin condition that does not require systemic therapy are exception to this criterion.
12. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent;
13. Live vaccine administration, within 30 days prior to the RFA;
14. Known allergy or hypersensitivity;
15. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with participation for the full duration of the trial;
16. Pregnancy and breastfeeding;
17. Tutelage or guardianship;
18. Patient refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult colorectal cancer patients, resectable or non-resectable liver metastases.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Plasma CD154 level dosage | at baseline
  Plasma CD154 level dosage realized by ELISA in patients with CRC liver metastases.
Plasma CD154 level dosage | at day 1
  Plasma CD154 level dosage realized by ELISA in patients with CRC liver metastases.
Plasma CD154 level dosage | at month 2
  Plasma CD154 level dosage realized by ELISA in patients with CRC liver metastases.

SECONDARY OUTCOMES:
Plasma CD154 level dosage in patients underwent surgery | at baseline, at day 1 and at month 2
  Plasma CD154 level dosage in patients underwent surgery for CRC.
Plasma CD154 level dosage evolution | at baseline, at day 1 and at month 2
  Plasma CD154 level dosage evolution.
Intraclass correlation of coefficient | at baseline, at day 1 and at month 2
  Intraclass correlation of coefficient to evaluate the feasibility and reliability of plasma CD154 level dosage in triplicate with CRC patients.
Rate of liver metastases relapses | at 1 year
  Liver metastases CRC relapses rate.
Clinical evolution parameters | at baseline, at day 1 and at month 2
  Clinical evolution parameters according to RECIST criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Robert MALAFOSSE, MD, Principal Investigator — Department of digestive surgery, Ambroise Paré Hospital, APHP; Cindy Neuzillet, MD, Study Director — Department of digestive surgery, Ambroise Paré Hospital, APHP
Locations (1):
- Department of digestive surgery, Ambroise Paré Hospital, APHP, Boulogne-Billancourt, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lemdani K, Mignet N, Boudy V, Seguin J, Oujagir E, Bawa O, Peschaud F, Emile JF, Capron C, Malafosse R. Local immunomodulation combined to radiofrequency ablation results in a complete cure of local and distant colorectal carcinoma. Oncoimmunology. 2019 Jan 10;8(3):1550342. doi: 10.1080/2162402X.2018.1550342. eCollection 2019. PMID 30723580
- [Background] Meier S, Stark R, Frentsch M, Thiel A. The influence of different stimulation conditions on the assessment of antigen-induced CD154 expression on CD4+ T cells. Cytometry A. 2008 Nov;73(11):1035-42. doi: 10.1002/cyto.a.20640. PMID 18785645
- [Background] Dymicka-Piekarska V, Korniluk A, Gryko M, Siergiejko E, Kemona H. Potential role of soluble CD40 ligand as inflammatory biomarker in colorectal cancer patients. Int J Biol Markers. 2014 Sep 30;29(3):e261-7. doi: 10.5301/jbm.5000083. PMID 24706377
- [Background] Tada N, Tsuno NH, Kawai K, Murono K, Nirei T, Ishihara S, Sunami E, Kitayama J, Watanabe T. Changes in the plasma levels of cytokines/chemokines for predicting the response to chemoradiation therapy in rectal cancer patients. Oncol Rep. 2014 Jan;31(1):463-71. doi: 10.3892/or.2013.2857. Epub 2013 Nov 19. PMID 24253593
- [Background] Zhao P, Fang WJ, Chai L, Ruan J, Zheng Y, Jiang WQ, Lin S, Zhou SH, Zhang ZL. The prognostic value of plasma soluble CD40 ligand levels in patients with nasopharyngeal carcinoma. Clin Chim Acta. 2015 Jul 20;447:66-70. doi: 10.1016/j.cca.2015.05.015. Epub 2015 May 29. PMID 26032866
- [Background] Allard MA, Bachet JB, Beauchet A, Julie C, Malafosse R, Penna C, Nordlinger B, Emile JF. Linear quantification of lymphoid infiltration of the tumor margin: a reproducible method, developed with colorectal cancer tissues, for assessing a highly variable prognostic factor. Diagn Pathol. 2012 Nov 13;7:156. doi: 10.1186/1746-1596-7-156. PMID 23148481